CLINICAL TRIAL: NCT07286084
Title: Effectiveness, Satisfaction, and Usability of Virtual Reality in the Management of Postoperative Pain in Patients Undergoing Knee Arthroplasty
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Francisco de Vitoria (Other)
Collaborators: University of Castilla-La Mancha (Other); Hospital Universitario del Sureste (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PI 94/25
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Knee Arthroplasty
Keywords: knee arthroplasty; postoperative pain; acute pain; virtual reality
MeSH Terms: conditions — Pain, Postoperative; Acute Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CONTROL (No Intervention): CONVENTIONAL TREATMENT
- EXPERIMENTAL (Experimental): VR GAMES
  Interventions: Device: VIRTUAL REALITY
- PLACEBO (Placebo Comparator): VR VIDEOS 360º
  Interventions: Device: VIRTUAL REALITY

INTERVENTIONS:
Device: VIRTUAL REALITY — Interactive VR Games: Participants use Meta Quest 3 head-mounted displays running a custom-developed VR application designed to elicit upper-limb and trunk movements. The application includes multiple structured scenarios:
  * Scenario 1 (Painting): Participants perform arm movements using handheld controllers to interact with a virtual painting environment.
  * Scenario 2 (Greenhouse): Participants move the arm to attract a butterfly, guide it toward a flower, and complete the assigned interaction task.
  * Scenario 3 (Aquarium): Participants perform bilateral arm movements to pop virtual bubbles.
  Immersive 360° Videos:Participants use Meta Quest 3 head-mounted displays to view immersive 360° relaxing videos (e.g., natural landscapes accompanied by calming background music).
  Arms: EXPERIMENTAL; PLACEBO

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of using virtual reality glasses to reduce the need for rescue analgesia in patients with acute postoperative pain after knee arthroplasty.

The main questions it aims to answer are:

* What is the impact of virtual reality use on postoperative pain perception as measured by the Visual Analogue Scale (VAS)?
* What potential adverse effects are associated with the use of virtual reality in the postoperative context?
* What is the level of satisfaction and acceptance of virtual reality as a complementary strategy for pain management?
* How does virtual reality influence quality of life and psychosocial variables in patients with acute postoperative pain after knee arthroplasty?

DETAILED DESCRIPTION:
A single-blind, randomized controlled trial will be conducted to compare gaming, 360° video viewing, and usual care interventions. Participants will be recruited from the prehabilitation clinic at Hospital del Sureste (Arganda del Rey), and the study will follow the CONSORT guidelines for clinical crossover and parallel trials.

Three experimental groups will be tested, with interventions performed at three different time points during hospitalization, each session lasting between 10 and 30 minutes. The gaming group will play video games, the control group will view 360° videos, and the usual care group will receive standard analgesia according to the protocol.

Outcome measures will be assessed at baseline (3 months before the intervention), during the intervention, and 1 month after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age, both sexes
* Scheduled unilateral knee arthroplasty
* Adequate cognitive and functional capacity to use virtual reality
* Signed informed consent

Exclusion Criteria:

* Neurological or psychiatric disorders (history of epilepsy, seizures, psychosis, schizophrenia, claustrophobia, tremor, rigidity)
* Significant visual or hearing impairments that hinder VR use
* Physical or motor limitations preventing the use of VR headsets or maintaining the required posture
* Score ≥4 on the 4AT delirium screening tool
* Pregnancy
* Recreational drug or alcohol use
* Inability to complete the intervention protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-12-27 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity (VAS) | Day 0 (day of intervention): pain measured at arrival to the ward and during three shifts (morning, afternoon, next-day morning), pre- and post conventional analgesia. If VR is used, pain is also measured immediately before and after each VR session.
  Pain intensity is assessed using a 100-mm Visual Analogue Scale (VAS), ranging from "no pain" (0 mm, left anchor) to "worst imaginable pain" (100 mm, right anchor). Higher scores indicate greater pain intensity.

SECONDARY OUTCOMES:
Sociodemographic variables | Baseline
  Age, weight, sex, and height recorded at enrollment
Analgesic medication use | From immediate postoperative period to 48 hours post-intervention.
  Analgesic administration (scheduled analgesia and rescue medication) is extracted from the hospital electronic medical record (Selene). Date and time of each dose are recorded to determine whether the intervention reduces short-term analgesic requirements.
Adverse events | Throughout the intervention period and up to 48 hours post-intervention.
  All adverse events reported by participants or investigators are documented and classified by intensity ("mild," "moderate," "severe") and by relatedness to the intervention ("none," "unlikely," "possible," "definite")
Satisfaction, Acceptability, and Perceived Safety (SEQ) | Immediately post-intervention
  The Suitability Evaluation Questionnaire (SEQ) assesses satisfaction, acceptability, usability, and perceived safety of the VR system. It includes 13 items rated from 1 ("not at all" or "very easy") to 5 ("very much" or "very difficult"), plus one open-ended question on discomfort
Health-Related Quality of Life (EQ-5D-5L) | Baseline and 1-month follow-up during outpatient visit
  The EQ-5D-5L assesses mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, each rated on a 5-level severity scale. Provides an individual health profile and utility index
Anxiety and depression (Goldberg Anxiety and Depression Scale) | Baseline and 1-month follow-up during outpatient visit
  The Goldberg Scale screens symptoms of anxiety and depression to explore changes associated with the intervention.
Physical Activity Level (IPAQ) | Baseline and 1-month follow-up during outpatient visit
  The International Physical Activity Questionnaire (IPAQ) assesses duration, frequency, and intensity of physical activity in the previous week, categorizing participants into low, moderate, or high activity levels.

IPD SHARING:
Plan to Share IPD: No